CLINICAL TRIAL: NCT01290224
Title: Scrambler Therapy for the Treatment of Chemotherapy Induced Peripheral Neuropathy: An Evaluation of a Sham Procedure and Phase II Trial
Brief Title: MC5-A Scrambler Therapy in Reducing Peripheral Neuropathy Caused by Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: MC10C8; NCI-2011-00109 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10-007874 (Other: Mayo Clinic IRB); MC10C8 (Other: Mayo Clinic Cancer Center)
Record Dates: First submitted 2011-02-01; First posted 2011-02-04 (Estimated); Results first posted 2014-03-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-01

CONDITIONS: Pain; Peripheral Neuropathy
MeSH Terms: conditions — Pain; Peripheral Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive Care (Experimental): See Detailed Description
  Interventions: Other: scrambler therapy; Procedure: sham intervention; Other: questionnaire administration

INTERVENTIONS:
Other: scrambler therapy — Undergo MC5-A therapy
  Other Names: TENPS; transcutaneous electromanipulation by nervous patterns scrambler therapy
Procedure: sham intervention — Undergo sham procedure
Other: questionnaire administration — Ancillary studies

SUMMARY:
RATIONALE: Scrambler therapy may help relieve pain from peripheral neuropathy caused by chemotherapy.

PURPOSE: This phase II trial is studying how well MC5-A scrambler therapy works in reducing peripheral neuropathy caused by chemotherapy

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To explore the feasibility of studying scrambler therapy versus a sham procedure for the alleviation of lower extremity chemotherapy induced peripheral neuropathy (CIPN).

SECONDARY OBJECTIVES:

I. To obtain prospective pilot experience with recommended scrambler therapy, with regards to treatment efficacy to determine effect size estimates, patient related outcome measurement tools that we use in this trial, tolerability, and analgesic use.

OUTLINE: Patients undergo a sham procedure on the back or scrambler therapy on both lower extremities for up to 30 minutes with the Calmare MC5-A device and cutaneous electrode patches applied above and below the area of pain on days 1 and 2. Patients continue scrambler therapy for 10 days in the absence of unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Received neurotoxic chemotherapy (including taxanes-such as paclitaxel or docetaxel, or platinum-based compounds such as carboplatin or cis-platinum or oxaliplatin, or vinca alkaloids such as vincristine, vinblastine, or vinorelbine, or proteosome inhibitors such as bortezomib); Note: this neurotoxic chemotherapy must have been completed more than 3 months prior to when they enter this trial
* Pain or symptoms of peripheral neuropathy in the feet of >= 1 month (30 days) duration attributed to chemotherapy-induced peripheral neuropathy, for which the patient wants intervention
* Participants have to relate that numbness, tingling or pain in their toes/feet was at least a four out of ten problem during the prior week, on a 0-10 scale where zero was no problem and ten was the worst possible problem
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) = 0, 1, or 2
* Life expectancy >= 3 months (90 days)
* Ability to complete questionnaire(s) by themselves or with assistance
* Provide informed written consent
* No change in scheduled analgesic agents for at least one week

Exclusion Criteria:

* Pregnant women
* CIPN troubles in the lower extremities more proximal to the mid calf
* Patients with implantable drug delivery systems, e.g. Medtronic Synchromed
* Patients with heart stents or metal implants such as pacemakers, automatic defibrillators, aneurysm clips, vena cava clips and skull plates; (metal implants for orthopedic repair, e.g. pins, clips, plates, cages, joint replacements are allowed as are central venous access devices)
* Patients with a history of myocardial infarction or ischemic heart disease within the past six months
* Patients with history of epilepsy, brain damage, use of anti-convulsants, symptomatic brain metastases
* Other identified causes of painful lower extremity paresthesias existing prior to chemotherapy (e.g., radiation or malignant plexopathy, lumbar or cervical radiculopathy, pre-existing peripheral neuropathy of another etiology: B12 deficiency, Acquired Immunodeficiency Syndrome [AIDS], monoclonal gammopathy, diabetes, heavy metal poisoning amyloidosis, syphilis, hyperthyroidism or hypothyroidism, inherited neuropathy, etc.)
* Skin conditions such as open sores that would prevent proper application of the electrodes
* Other medical or other condition(s) that in the opinion of the investigators might compromise the objectives of the study
* Prior treatment with Calmare MC-5A therapy for any reason or knowledge of application procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Loprinzi, M.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ten (10) participants were recruited at Mayo Clinic between February 2011 and April 2011. All 10 participants have completed sham procedure (day 1) and proceed to scrambler treatment (day 2 to 11).
Period: Overall Study
Arm/Group | Sham Procedure + Scrambler Treatment
Started | 10
Completed | 5
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Refused Further Treatment | 4

BASELINE CHARACTERISTICS:
Arm/Group | Sham Procedure + Scrambler Treatment
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Number of neurotoxic agents exposed to [Number; unit: participants]
  Single Agent | 7
  Multiple Agents | 3
Duration of pain symptoms at baseline [Number; unit: participants]
  <=6 months | 10
  >6 months | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Have at Least a 50% Reduction (i.e., Success) in at Least 1 of the First 12 Chemotherapy Induced Peripheral Neuropathy (CIPN) Measurement Questions in the Pre/Post Therapy Questionnaire
Description: CIPN measurement items score range: 0 (none) to 10 (as bad as can be). The questions assessed the intensity of numbness, tingling, or pain in toes or feet that patients have had right now, at its worst over the past 24 hours, and on average over the past 24 hours.
Time Frame: On days 1 and 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Sham Procedure + Scrambler Treatment
Number analyzed (Participants) | 10
Percentage of Participants
  Sham Procedure | 60
  Scrambler Therapy | 50
Statistical Analysis 1: Comparison: Sham Procedure + Scrambler Treatment; McNemar's test was used to test for a difference between Scrambler and Sham procedure in their success rate; Test type: Non-Inferiority or Equivalence — A one-sided McNemar's test of the primary endpoint with 10 patients will have 86% power at 5% Type I error rate to detect a 60% difference in the percentage of at least 50% reduction in the scrambler and sham procedure, based on the assumption that the proportion of discordant pairs is at 70%; p = 0.7630, McNemar

2. Secondary Outcome: Average Change of CIPN Symptoms Between Sham Procedure and Scrambler Therapy as Measured by Each Individual Question
Description: The 12 CIPN symptoms individual question range: 0 (none) to 10 (as bad as can be). The questions assessed the intensity of numbness, tingling, or pain in toes or feet that patients have had right now (RN), at its worst over the past 24 hours (WP24H), and on average over the past 24 hours (AvgP24H). Averaged change between day 1 and day 2 across 10 patients was calculated.
Time Frame: On days 1 and 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Procedure (Day 1 ) | Scrambler Therapy (Day 2)
Number analyzed (Participants) | 10 | 10
units on a scale
  Numbness, tingling, or pain in toes/feet RN | -1 (1.49) | -0.2 (1.62)
  Numbness in toes/feet RN | -0.8 (1.40) | -0.5 (0.85)
  Tingling in toes/feet RN | -0.8 (1.32) | -0.8 (1.55)
  Pain in toes/feet RN | 0 (1.41) | 0.1 (1.60)
  Numbness, tingling, or pain in toes/feet at WP24H | -0.7 (1.25) | 0 (0.94)
  Numbness in toes/feet at WP24H | -0.6 (1.35) | -0.7 (0.82)
  Tingling in toes/feet at WP24H | -0.7 (0.95) | -0.2 (0.42)
  Pain in toes/feet at WP24H | 0.1 (0.74) | 0.2 (1.40)
  Numbness, tingling, or pain in toes/feet AvgP24H | -0.4 (0.70) | -0.6 (2.27)
  Numbness in toes/feet AvgP24H | -0.6 (1.17) | -0.8 (1.32)
  Tingling in toes/feet AvgP24H | -0.1 (1.45) | -0.2 (1.14)
  Pain in toes/feet AvgP24H | -0.3 (1.77) | -0.2 (1.03)

3. Secondary Outcome: Percentage of Reduction at Days 10 From Day 1 in Each of the 12 CIPN Measurement Questions in the Daily Therapy Questionnaire
Description: The 12 CIPN symptoms individual question range: 0 (none) to 10 (as bad as can be). The questions assessed the intensity of numbness, tingling, or pain in toes or feet that patients have had right now (RN), at its worst over the past 24 hours (WP24H), and on average over the past 24 hours (AvgP24H).
Time Frame: Day 1 and Day 10
Measure: Mean (Standard Deviation); unit: percentage of reduction in symptom
Arm/Group | Sham Procedure + Scrambler Treatment
Number analyzed (Participants) | 10
percentage of reduction in symptom
  Numbness, tingling, or pain in toes/feet RN | 43.5 (41.7)
  Numbness in toes/feet RN | 46.7 (36.3)
  Tingling in toes/feet RN | 37.8 (57.7)
  Pain in toes/feet RN | 13.4 (89.3)
  Numbness, tingling, or pain in toes/feet at WP24H | 12.8 (52.0)
  Numbness in toes/feet at WP24H | 40.6 (37.5)
  Tingling in toes/feet at WP24H | 50.6 (47.6)
  Pain in toes/feet at WP24H (Worsen) | -8.3 (99.1)
  Numbness, tingling or pain in toes/feet AvgP24H | 23.5 (27.9)
  Numbness in toes/feet AvgP24H | 45.2 (32.2)
  Tingling in toes/feet AvgP24H | 48.4 (46.8)
  Pain in toes/feet AvgP24H | 26.6 (70.8)

4. Secondary Outcome: Percentage of Reduction at Weeks 10 From Week 1 in CIPN Symptoms as Measured by the North Central Cancer Treatment Group (NCCTG) Peripheral Neuropathy Question
Description: The NCCTG peripheral neuropathy question range: 0 (No numbness or tingling or pain in fingers and/or toes) to 10 (Numbness, tingling or pain in fingers and/pr toes as bad as you can imagine). The question assessed the intensity of numbness, tingling or pain in toes or feet in the past week.
Time Frame: Week 1 and Week 10
Measure: Mean (Standard Deviation); unit: percentage of reduction in symptom
Arm/Group | Sham Procedure + Scrambler Treatment
Number analyzed (Participants) | 10
percentage of reduction in symptom | 3.2 (38.6)

5. Secondary Outcome: Percent Change From Day 1 at Week 10 in CIPN Symptom Bother as Measured by 8 CIPN Symptom Questions
Description: The intensity of symptom was measured in a likert scale: none at all (0), a little bit (1), quite a bit (2) and very much (3). Percent change from day 1 at week 10 for each patient was calculated and average of percentage was reported.
Time Frame: Day 1 and Week 10
Measure: Mean (Standard Deviation); unit: percentage of a scale
Arm/Group | Sham Procedure + Scrambler Treatment
Number analyzed (Participants) | 10
percentage of a scale
  Tingling in toes/feet | 42.9 (45.0)
  Numbness in toes/feet | -25.0 (46.3)
  Shooting/burning in toes/feet | -10.0 (89.4)
  Problems standing/walking | 21.4 (39.3)
  Cramps in toes/feet | 50.0 (44.7)
  Difficulty walking | 16.7 (25.8)
  Difficulty with stairs | 20.0 (27.4)
  Difficulty using car foot pedals | 20.0 (44.7)

6. Secondary Outcome: Toxicity (Other Than CIPN) Profile Associated With Scrambler Therapy as Measured by Common Terminology Criteria for Adverse Events (CTCAE) 4.0
Description: CTCAE Grading: Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening, Grade 5=Death.
Time Frame: Day 1 to Day 10
Measure: Number; unit: participants
Arm/Group | Sham Procedure + Scrambler Treatment
Number analyzed (Participants) | 10
participants
  Grade 1, 2 | 1
  Grade 3, 4, 5 | 0

7. Secondary Outcome: Analgesic Use Over Time
Time Frame: On days 1-11 and for 10 weeks after therapy
Measure: Number; unit: participants
Arm/Group | Sham Procedure + Scrambler Treatment
Number analyzed (Participants) | 10
participants
  Tylenol | 3
  Ibuprofen | 3
  Cymbalta | 1
  Lyrica | 1
  Tramadol | 1
  Gabapentin | 1
  Acetaminophen | 2
  Oxycontin | 1
  Oxycodone | 1

ADVERSE EVENTS:
Time Frame: 11 days
Description: NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 was utilized for AE reporting. The adverse event: musculoskeletal/connective tissue disorder was reported on day 3, which is during the scrambler treatment period.
Arm/Group | Sham Procedure + Scrambler Treatment
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Procedure + Scrambler Treatment (N=10)
Musculoskeletal/connective tissue disorder - achiness, fatigue and heaviness in bilateral lower legs (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No